CLINICAL TRIAL: NCT04974216
Title: Phase II, Open-Label Study Evaluating Efficacy of Tafasitamab and Lenalinomide Associated to Rituximab in Frontline Diffuse Large B-Cell Lymphoma Patients of 80 y/o or Older
Brief Title: Study of Tafasitamab and Lenalinomide Associated to Rituximab in Frontline Diffuse Large B-Cell Lymphoma Patients of 80 y/o or Older
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VERLen
Record Dates: First submitted 2021-07-13; First posted 2021-07-23 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: DLBCL
MeSH Terms: interventions — tafasitamab; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-Lena-Tafa (Experimental): 12 cycles of 28 days. From C1 to C6 : rituximab + tafasitamab + lenalidomide and from C7 to C12: tafasitamab and lenalidomide
  Patients with Progressive Disease or Stable Disease after 3 cycles should start a conventional chemotherapy (rituximab + cyclophosphamide + adriamycine + vincristine + prednisone R-miniCHOP) at Investigator's discretion according to local practices
  Interventions: Drug: Tafasitamab; Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Tafasitamab — Administration : IV at 12mg/Kg C1 to C3: D1, D8, D15, D22 C4 to C6: D1, D15 C7 to C12: D1
  Other Names: MOR208
Drug: Lenalidomide — Oral administration: hard capsule C1 to C6: 20mg/day C7 to C12: 15mg/day
Drug: Rituximab — Administration: IV at 375mg/m2 C1 to C6: D1

SUMMARY:
This study evaluate the efficacy of Tafasitamab and Lenalinomide associated to Rituximab in elderly patients with frontline Diffuse Large B-Cell Lymphoma as assessed by the Overall Response Rate (ORR) after 3 cycles of treatment according to Lugano Response Criteria.

DETAILED DESCRIPTION:
This study is an open-label, multi-centric, phase II study designed to evaluate the efficacy of Tafasitamab and Lenalinomide associated to Rituximab in elderly patients with frontline Diffuse Large B-Cell Lymphoma as assessed by the Overall Response Rate (ORR) after 3 cycles of treatment according to Lugano Response Criteria.

After a screening phase, eligible patients will be enrolled and start the prephase treatment with vincristine and prednisone before day 1 of cycle 1 of the experimental drugs.

Patients with Progressive Disease or Stable Disease after 3 cycles should start a conventional chemotherapy (R-miniCHOP) at Investigator's discretion and will remain in the study.

ELIGIBILITY:
Inclusion Criteria:

2.Patient with histologically proven CD20+ diffuse large B-cell lymphoma (DLBCL) (WHO classification 2017) including all clinical subtypes (primary mediastinal, intravascular, etc…), with all International Prognostic Index (IPI). May also be enrolled the following malignancies:

* De Novo transformed DLBCL from low grade lymphoma (Follicular, other...) and DLBCL associated with some small cell infiltration in bone marrow or lymph node.
* High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements
* High-grade B-cell lymphoma, Not Otherwise Specified (NOS)
* Follicular lymphoma grade 3B 3.Positron-Emission Tomography (PET)-positive disease 4.Previously untreated high-grade B-cell lymphoma 5.Aged ≥ 80 years old at the time of signing the informed consent form (ICF) 6.Ann Arbor stage I, II, III or IV 7.Eastern Cooperative Oncology Group (ECO)G performance status ≤ 2 8.With a minimum life expectancy of 3 months 9.Male patients must practice complete abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for 4 months following study drug discontinuation, even if they have undergone a successful vasectomy 10. Patients should be able to receive R-miniCHOP regimen (left ventricular ejection fraction > 50% and good general condition, according to investigator's judgment) 11. Patients should be able to receive adequate prophylaxis and/or therapy for thromboembolic events (aspirin or low molecular weight heparin) 12. Patient covered by any social security system (France)

Exclusion Criteria:

1. Any other histological type of lymphoma, Burkitt included
2. Any history of treated or non-treated Small-B cell lymphoma prior Aggressive B Cell lymphoma diagnosis
3. Central nervous system or meningeal involvement by lymphoma
4. Any serious active disease (according to the investigator's decision)
5. Poor renal function (calculated Cockcroft-Gault creatinine clearance < 30 ml/min)
6. Poor hepatic function (total bilirubin level >30 μmol/l, transaminases >2.5 upper normal limits) unless these abnormalities are related to lymphoma
7. Poor bone marrow reserve as defined by neutrophils <1.5 G/l or platelets <100 G/l, unless related to bone marrow infiltration by lymphoma cells (Bone Marrow Aspiration will be mandatory in case of severe cytopenias prior inclusion)
8. Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma. Patients previously diagnosed with prostate cancer are eligible if (1) their disease was T1-T2a, N0, M0, with a Gleason score ≤7, and a prostate specific antigen (PSA) ≤10 ng/mL prior to initial therapy, (2) they had definitive curative therapy (i.e., prostatectomy or radiotherapy) 2 years before Day 1 of Cycle 1, and (3) at a minimum 2 years following therapy they had no clinical evidence of prostate cancer, and their PSA was undetectable if they underwent prostatectomy or <1 ng/mL if they did not undergo prostatectomy
9. Treatment with any investigational drug within 30 days prior to prephase treatment and during the study
10. Known HIV, active Hepatitis C Virus (HCV) infection or positive Hepatitis B Virus (HBV) test within 4 weeks before enrollment (except after hepatitis B vaccination or for patients who are HBs Ag negative, anti-HBs positive and/or anti-HBc positive but viral DNA negative)
11. Prior treatment with anti-CD20/anti-CD19 monoclonal antibody or alemtuzumab within 3 months prior to prephase treatment
12. Prior ≥ Grade 3 allergic reaction/hypersensitivity to thalidomide
13. Contra-indication to highly dosed glucocorticoid (60 mg/m2/d)
14. Neuropathy ≥ Grade 2 or painful
15. Patient deprived of his/her liberty by a judicial or administrative decision
16. Adult patient under legal protection

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) by local assessment | 3 months (3 cycles of 28 days)
  LOCAL ASSESSMENT : Complete Metabolic Response + Partial Metabolic Response based according to Lugano Response Criteria

SECONDARY OUTCOMES:
Number of Serious Adverse Events (SAE) of patients treated with lenalidomide and tafasitamab | 13 months
Number of SAE of patients who switched to RminiCHOP | 7 months
Progression free survival (PFS) | 2 years
Overall survival (OS) | 2 years
Overall Response Rate (ORR) by central assessment | 3 months (3 cycles of 28 days)
  CENTRAL ASSESSMENT : Complete Metabolic Response + Partial Metabolic Response based according to Lugano Response Criteria
Complete Metabolic Response (CMR) by local assessment | 3 months (3 cycles of 28 days)
  LOCAL ASSESSMENT
Complete Metabolic Response (CMR) by central assessment | 3 months (3 cycles of 28 days)
  CENTRAL ASSESSMENT
Complete Metabolic Response (CMR) by local assessment | 6 months (6 cycles of 28 days)
  LOCAL ASSESSMENT
Complete Metabolic Response (CMR) by central assessment | 6 months (6 cycles of 28 days)
  CENTRAL ASSESSMENT
Complete Metabolic Response (CMR) by local assessment | 12 months (12 cycles of 28 days = end of treatment)
  LOCAL ASSESSMENT
Complete Metabolic Response (CMR) by central assessment | 12 months (12 cycles of 28 days = end of treatment)
  CENTRAL ASSESSMENT
Overall Response Rate (ORR) by local assessment | 6 months (6 cycles of 28 days)
  LOCAL ASSESSMENT : Complete Metabolic Response + Partial Metabolic Response based according to Lugano Response Criteria
Overall Response Rate (ORR) by central assessment | 6 months (6 cycles of 28 days)
  CENTRAL ASSESSMENT : Complete Metabolic Response + Partial Metabolic Response based according to Lugano Response Criteria
Overall Response Rate (ORR) by local assessment | 12 months (12 cycles of 28 days = end of treatment)
  LOCAL ASSESSMENT : Complete Metabolic Response + Partial Metabolic Response based according to Lugano Response Criteria
Overall Response Rate (ORR) by central assessment | 12 months (12 cycles of 28 days = end of treatment)
  CENTRAL ASSESSMENT : Complete Metabolic Response + Partial Metabolic Response based according to Lugano Response Criteria
Progression free survival (PFS) of patients who switched to RminiCHOP | 3 years
Overall survival (OS) of patients who switched to RminiCHOP | 3 years

CONTACTS AND LOCATIONS:
Locations (15):
- Belgium (3):
  - Clinique Universitaire Saint LUC, Brussels
  - CHU de Liège, Liège
  - CHRU Mont Godinne, Yvoir
- France (12):
  - CHU de Bordeaux - Hôpital Haut Lévêque, Bordeaux
  - Institut Bergonié - Bordeaux, Bordeaux
  - CH Saint Vincent de Paul, Lille
  - CHRU de LILLE - Claude Huriez, Lille
  - Chu de Limoges - Hopital Dupuytren, Limoges
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - APHP - Hôpital Saint Louis, Paris
  - Centre Henri Becquerel, Rouen
  - Centre René Huguenin - Institut Curie, Saint-Cloud
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - CHU Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No